CLINICAL TRIAL: NCT01944306
Title: Prenatal Growth Programs Oral Contraceptive Metabolism and Effectiveness
Brief Title: Obesity and Oral Contraceptive Failure
Status: Terminated | Type: Observational
Why Stopped: Due to lack of funds, the study has been terminated upon recruiting less than desired number of subjects
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00009569; 2K12HD043488-11 (NIH)
Record Dates: First submitted 2013-09-10; First posted 2013-09-17 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Contraception; Fetal Growth Retardation; Infant, Small for Gestational Age; Obesity
Keywords: Pharmacokinetics; Pharmacology, Clinical; Drug Efficacy; Drug Failure; Contraceptive Agents
MeSH Terms: conditions — Fetal Growth Retardation; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Plasma, and Urine will be collected for the analaysis of drug levels and genotyping of various genes that could explain pharmacokinetics of oral contraceptives.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Low birth-weight, obese
- Low birth-weight, normal body weight
- Normal birth-weight, obese
- Normal birth-weight, normal body weight

SUMMARY:
Contraceptive failure is the primary cause of unintended pregnancy in the United States. With obesity rates at epidemic proportions, any association between obesity and strategies that prevent undesired pregnancies constitutes a significant public health and economic concern. Evidence from recent epidemiological studies and our preliminary data (sub-therapeutic levels of steroid hormones due to drug clearance and half-life) suggest that obesity reduces oral contraceptive efficacy. Furthermore, preliminary analysis suggested that a sub-group of obese women, defined by their own birth weight, are at higher risk of contraceptive failure. Further studies are necessary to investigate whether birth weight, a surrogate marker of in utero growth restriction, is a useful diagnostic marker for the identification of women prone to contraceptive failure. Such an understanding is critical to finding a contraceptive strategy with better efficacy for these women.

The overall goal of this project is to test pharmacokinetics of oral contraceptive agents in obese women with low birth weight and compare to obese women with normal birth weight. The main hypothesis for this proposal is that an adverse in utero environment programs the expression and function of enzymes and transporters that underlie pharmacokinetics of oral contraceptives, and leads to contraceptive failure.

Reproductive-aged, ovulatory women of obese BMI >30 kg/m2 with normal birth weight (5.5-8 lbs; n=10) and low birth weight (<5.5 lbs; n=10), will be placed on oral contraceptives for 1 month. At several key time points, synthetic steroid pharmacokinetics, gonadotropins (luteinizing hormone, follicle-stimulating hormone) and ovarian hormone levels (estradiol, progesterone) will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 35.
* single progesterone level of 3 ng/mL or greater during the luteal phase (days 18 to 25) in the menstrual cycle prior to dosing with oral contraceptives.

Exclusion Criteria:

* absolute/relative contraindications to ethinyl estradiol and levonorgestrel.
* impaired liver function.
* history of deep venous thrombosis.
* hypertension (> 140/90).
* diabetes with vascular changes.
* migraines with aura or neurological changes.
* history of myocardial infarction, pulmonary embolus, stroke or breast cancer.
* anemia (hematocrit < 36%).
* actively seeking or involved in a weight loss program (must be weight stable)
* pregnancy, breastfeeding, or seeking pregnancy.
* diagnosis of Polycystic Ovarian Syndrome.
* recent (4 week) use of hormonal contraceptives (patch or ring included), intrauterine, or implantable hormonal contraception.
* DepoProvera use within six months.
* current use of drugs that interfere with metabolism of sex steroids.
* smokers.
* uncontrolled thyroid dysfunction.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Reproductive-aged, ovulatory women seeking to initiate contraception with combined oral contraceptives will be recruited from the female population of the Portland, OR area. Subjects must have access to their birth weight record. Enrollment will be confined to women who have not used a hormonal contraceptive method for 30 days or more prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Measure pharmacokinetic parameters of oral contraceptives including drug clearance. | on day 21 of oral contraceptive use
  Serum concentration-time data for each subject will be analyzed using a non-compartmental model assumption. Serum concentrations below the lower limit of quantitation (LLOQ) at the beginning and end of the profile will be set to zero. Serum concentration-time profiles will be summarized using descriptive statistics and graphical display. Student t-tests will be used to test whether the average values of each of the pharmacokinetic parameters, including free concentrations, differ between the four groups of women.

SECONDARY OUTCOMES:
Measure levels of gonadotropins and ovarian hormones | Days 21-25 of oral contraceptive use
  To compare gonadotopin levels, average leutinizing hormone and follicle stimulating hormone levels measured for days 21-25 will be calculated. In addition, the follicle stimulating hormone/leutinizing hormone ratio will be calculated at each time point. The average levels of these measures will then be compared between the four groups of women using a student's t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Cherala, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Edelman AB, Carlson NE, Cherala G, Munar MY, Stouffer RL, Cameron JL, Stanczyk FZ, Jensen JT. Impact of obesity on oral contraceptive pharmacokinetics and hypothalamic-pituitary-ovarian activity. Contraception. 2009 Aug;80(2):119-27. doi: 10.1016/j.contraception.2009.04.011. Epub 2009 Jun 4. PMID 19631786
- [Background] Cherala G, Thornburg K, Edelman A. Birthweight and cytochrome P4503A4/5 activity in obese women. Br J Clin Pharmacol. 2013 Jan;75(1):275-6. doi: 10.1111/j.1365-2125.2012.04309.x. No abstract available. PMID 22534035
- [Background] Edelman AB, Cherala G, Munar MY, Dubois B, McInnis M, Stanczyk FZ, Jensen JT. Prolonged monitoring of ethinyl estradiol and levonorgestrel levels confirms an altered pharmacokinetic profile in obese oral contraceptives users. Contraception. 2013 Feb;87(2):220-6. doi: 10.1016/j.contraception.2012.10.008. Epub 2012 Nov 12. PMID 23153898
- [Background] Edelman A, Cherala G, Lim JY, Jensen JT. Contraceptive failures in overweight and obese combined hormonal contraceptive users. Obstet Gynecol. 2013 Jul;122(1):158-159. doi: 10.1097/AOG.0b013e3182995811. No abstract available. PMID 23787930